CLINICAL TRIAL: NCT06570031
Title: ONO-4578-06: Phase I , Open-label, Non-blind, First-line Endocrine Therapy With ONO-4578 and Standard Treatment Letrozole and CDK4/6 Inhibitors (Palbociclib or Abemaciclib) in Patients With Metastatic or Recurrent Postmenopausal Hormone Receptor-positive HER2-negative Breast Cancer
Brief Title: ONO-4578-06:Phase I Study of ONO-4578 and Letrozole Plus CDK4 /6 Inhibitors in Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-06
Record Dates: First submitted 2024-07-31; First posted 2024-08-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hormone Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: Breast Cancer; Hormone Receptor-positive; HER2-negative; Metastatic; Recurrent
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Letrozole; palbociclib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ONO-4578 + letrozole + palbociclib (Experimental)
  Interventions: Drug: ONO-4578; Drug: letrozole; Drug: Palbociclib
- ONO-4578 + letrozole + abemaciclib (Experimental)
  Interventions: Drug: ONO-4578; Drug: letrozole; Drug: abemaciclib

INTERVENTIONS:
Drug: ONO-4578 — Specified dose on specified days
Drug: letrozole — Specified dose on specified days
Drug: Palbociclib — Specified dose on specified days
  Arms: ONO-4578 + letrozole + palbociclib
Drug: abemaciclib — Specified dose on specified days
  Arms: ONO-4578 + letrozole + abemaciclib

SUMMARY:
This is a multicenter, open-label, non-controlled, phase I study to investigate the tolerability and safety of ONO-4578 used in combination with standard-of-care letrozole and a CDK4/6 inhibitor (palbociclib or Abemaciclib) as first-line endocrine therapy in postmenopausal patients with metastatic or recurrent hormone receptor-positive, HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with postmenopausal metastatic or recurrent breast cancer
2. Patients with ECOG Performance Status 0 to 1
3. ER-positive, PgR-positive and HER2-negative patients

Exclusion Criteria:

1. Patients are unable to swallow oral medications
2. Patients with severe complication

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 4 year
Serious adverse events | Through study completion, an average of 4 year
Dose-limiting toxicity (Tolerability Confirmation part only) | 28 days
Laboratory abnormality profile of Drugs as measured by incidence and severity of clinical laboratory abnormalities | Through study completion, an average of 4 year
Body temperature | Through study completion, an average of 4 year
Pulse rate | Through study completion, an average of 4 year
Systolic/diastolic blood pressure | Through study completion, an average of 4 year
Saturation of Percutaneous Oxygen (SpO2) | Through study completion, an average of 4 year
Weight | Through study completion, an average of 4 year
Eastern Cooperative Oncology Group Performance Status | Through study completion, an average of 4 year
Chest X-ray | Through study completion, an average of 4 year
CT scan | Through study completion, an average of 4 year
12-lead electrocardiography (Heart rate) | Through study completion, an average of 4 year
12-lead electrocardiography (PR interval) | Through study completion, an average of 4 year
12-lead electrocardiography (RR interval) | Through study completion, an average of 4 year
12-lead electrocardiography (QRS width) | Through study completion, an average of 4 year
12-lead electrocardiography (QT interval) | Through study completion, an average of 4 year

SECONDARY OUTCOMES:
Overall response rate (ORR) | Through study completion, an average of 4 year
Disease control rate (DCR) | Through study completion, an average of 4 year
Clinical benefit rate (CBR) | Through study completion, an average of 4 year
Overall survival (OS) | Through study completion, an average of 4 year
Progression-free survival (PFS) | Through study completion, an average of 4 year
Duration of response (DOR) | Through study completion, an average of 4 year
Time to response (TTR) | Through study completion, an average of 4 year
Best overall response (BOR) | Through study completion, an average of 4 year
Percent change in the sum of diameters of target lesions | Through study completion, an average of 4 year
Maximum percent change in the sum of diameters of target lesions | Through study completion, an average of 4 year
Changes in tumor markers | Through study completion, an average of 4 year
Plasma ONO-4578 concentration | Through study completion, an average of 4 year

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (13):
- Japan (13):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - Saitama Cancer Center, Shinden, Saitama
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No